CLINICAL TRIAL: NCT03679702
Title: A Viveve Experience Normalizes Untreated Selective Serotonin Reuptake Inhibitor (SSRI) Sexuality Syndrome
Acronym: VENUSSSS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Michael Krychman, MD (Other)
Collaborators: Viveve Inc. (Industry)
Responsible Party: Sponsor-Investigator, Michael Krychman, MD, Michael Krychman, MD, Southern California Center for Sexual Health and Survivorship Medicine
Organization: Southern California Center for Sexual Health and Survivorship Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VI-ISRP-034
Record Dates: First submitted 2018-09-19; First posted 2018-09-20 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Sexual Dysfunction
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Active treatment (Other)
  Interventions: Device: Viveve System

INTERVENTIONS:
Device: Viveve System — Radiofrequency device utilized in general surgical procedures for electrocoagulation and hemostasis.

SUMMARY:
A pilot study to investigate non-surgical treatment for women who suffer from sexual complaints secondary to SSRI Sexuality Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Currently using SSRI for 3 months at a stable dose

Exclusion Criteria:

* Pregnant, currently breastfeeding, or breast-fed within the last 6 months
* Has any implantable electrical device that could potentially be affected by use of radiofrequency.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-12-15 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety - Adverse Events | baseline to 6 month
  safety of treatment of female sexual dysfunction secondary to SSRI sexuality syndrome

SECONDARY OUTCOMES:
Female Sexual Function Index (FSFI) | baseline to 3 and 6 months
  Female Sexual Function Index total score (Minimum: 2.0) (Maximum: 36), Higher scores are better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Southern California Center for Sexual Health and Survivorship Medicine, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No